CLINICAL TRIAL: NCT03771924
Title: Postprandial Response of Individuals to Dietary Inorganic Phosphate- a Randomized Trial
Brief Title: Postprandial Response of Individuals to Dietary Inorganic Phosphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Ulf Schlegelmilch, Study Coordinator, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BMBF WP2A3
Record Dates: First submitted 2018-11-07; First posted 2018-12-11 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: inorganic phosphate; postprandial response; fibroblast growth factor-23; health individuals
MeSH Terms: interventions — Phosphates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inorganic phosphate (Experimental): Experimental intervention:
  Single dose of orally administered 700 mg inorganic phosphate as sodium phosphate in combination with a standardized meal and blood sampling
  Interventions: Dietary Supplement: inorganic phosphate
- Placebo (Placebo Comparator): Single dose of Sodium chloride in combination with a standardized meal and blood sampling
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: inorganic phosphate — Sodium phosphate
  Arms: inorganic phosphate
Dietary Supplement: placebo — Sodium chlorid
  Arms: Placebo

SUMMARY:
The study aims to compare the postprandial response of plasma phosphate and cardiometabolic relevant factors to phosphate intake in defined diet(s).

DETAILED DESCRIPTION:
It is a monocentric, controlled intervention trial. The study will be carried out in cross-over design. This design was chosen because of a moderately strong individual metabolic response to the test meal.

Two interventions are planned in which the subjects will receive a test meal with phosphate supplement or with placebo in random order on 2 days. Subjects will be randomized to one of the 2 treatment arms.

On the two intervention days (T1 and T2), the subjects are placed a venous indwelling cannula. Immediately after the first blood sample the subjects take the fat and carbohydrate-rich test meal along with 700 mg of phosphorus or a placebo, both in the form of capsules. Phosphorus is administered as sodium phosphate . The placebo used is sodium chloride with equivalent amounts of sodium. The filler should be silica and mannitol. The capsules are made of hard gelatin and dissolve in about 10 minutes. The capsules are taken with 300 ml of water. The verum and placebo capsules are produced by the central pharmacy of the University Hospital.

The test meal consists of a pasta dish with oily tomato sauce. It is freshly prepared by the study staff and packaged airtight in individual portions before being handed out to the subjects. The test meal should be consumed within 10 - 12 minutes. The time is documented by the study staff. The next blood sample is taken immediately after the end of consumption (time 0), all other 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420 and 480 minutes thereafter. All blood samples are taken in a lying position. The first 3 hours after eating the test meal the subjects should spend reclining. In the following 5 hours subjects are free to move in the study center with each patient taking a recumbent position 10 minutes before the next blood draw. Immediately before all blood samples are taken the measurement of blood pressure and pulse is provided for which the opposite arm is to be used. Furthermore the collection of urine samples is provided every hour. Subjects are encouraged to take 200 ml of water every hour on the intervention day. At the end of the intervention, a snack will be provided.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age between 18 and 60 years
* informed consent
* body mass index between 18,5 up to 29,9 kg/m2
* anamnesis without diagnostic findings

Exclusion Criteria:

* Participants with epidermal growth factor receptor (eGFR) < 90 ml/min and chronic kidney disease
* Subjects suffering from vitamin D-deficiency (plasma 25(OH)D < 30 nmol/l)
* Pregnancy or lactation
* Subjects with any acute or chronic diseases (infection, tumor, cardiovascular diseases, respiratory diseases, inflammatory diseases), gastrointestinal diseases, diabetes mellitus type 1 and 2, bone diseases, diseases of the parathyroid gland
* Use of medication
* Use of dietary supplements (minerals)
* Relevant food allergies (wheat protein, tomatoes)
* Weight reduction
* Smokers
* Blood donor in the last 3 months
* Participation in another intervention study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Postprandial change of plasma phosphate concentration from baseline (0 minute) until 480 minutes | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels of plasma phosphate concentration

SECONDARY OUTCOMES:
Postprandial course of the plasma concentration of: electrolytes (calcium, sodium, potassium, magnesium) | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of the plasma concentration of: phosphate status markers (c-terminal and intact FGF23, parathormone, soluble Klotho (sKlotho), calcitriol) | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of plasma concentration of: cardiovascular risk marker glucose | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of plasma concentration of: cardiovascular risk marker insulin | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of plasma concentration of: cardiovascular risk marker triglycerides | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of plasma concentration of: cardiovascular risk marker cholesterol | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Postprandial course of concentration of: calcification markers dephosphorylated, noncarboxylated matrix Gla protein (dp-ucMGP), fetuin A, osteocalcin, osteoprotegerin) Inflammatory markers (hsCRP and inflammatory cytokines, especially interleukin (IL-1β) | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
Activation of NLRP3-inflammasome components (ASC, caspase-1) in isolated peripheral blood monocytes (PBMC) and granulocytes under basal conditions and after stimulation | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels
systolic and diastolic blood pressures | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  time course: measurement of blood pressure in mm Hg
heart rate | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  time course: measurement of heart rate in beats per minute
Postprandial course of urine concentrations of electrolytes (phosphate, sodium, potassium, calcium, magnesium) and creatinine | 0,15,30,45,60,90,120,180,240,300, 360, 420 and 480 minutes after ingestion of testmeal rich in carbohydrates and fat
  Impact of inorganic phosphate on the postprandial levels

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Stangl, Prof.Dr., Study Director — MLU, Institut für Agrar-und Ernährungswissenschaften
Locations (1):
- Martin-Luther-University Institute of Agriculture and Nutritional Science, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Derived] Nier A, Ulrich C, Volk C, Wolffgang MC, Brandsch C, Wensch-Dorendorf M, Girndt M, Stangl GI. Effects of a single phosphate-enriched test meal on inflammasome activity and postprandial inflammatory markers in healthy subjects. Eur J Nutr. 2024 Apr;63(3):797-807. doi: 10.1007/s00394-023-03306-6. Epub 2024 Jan 4. PMID 38175251